CLINICAL TRIAL: NCT04762836
Title: Manipulating NMDA-dependent Learning to Alter Nocebo Effects: A Pharmacological fMRI Study on Pain
Brief Title: Pain, Learning, and Nocebo
Acronym: PIPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Leiden University (Other)
Responsible Party: Principal Investigator, AWMEvers, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL66693.058.18
Record Dates: First submitted 2020-12-13; First posted 2021-02-21 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain; Pain Syndrome
Keywords: Nocebo; Pain; BOLD; fMRI; Conditioning
MeSH Terms: conditions — Chronic Pain; Somatoform Disorders; Pain | interventions — Cycloserine; Extinction, Biological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented learning (Experimental): Conditioning and extinction of a nocebo response to the activation of a sham electrode, controlled within subjects. All participants in this arm receive a double-blind oral dose of DCS two hours prior to conditioning and fMRI
  Interventions: Drug: D-cycloserine; Behavioral: Conditioning; Behavioral: Extinction; Other: fMRI
- Baseline learning (Placebo Comparator): Conditioning and extinction of a nocebo response to the activation of a sham electrode, controlled within subjects. All participants in this arm receive a double-blind oral dose of placebo two hours prior to conditioning and fMRI
  Interventions: Behavioral: Conditioning; Behavioral: Extinction; Other: fMRI; Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — Antibiotic medication that augments the function of NMDA-receptors
  Other Names: DCS
  Arms: Augmented learning
Behavioral: Conditioning — During nocebo acquisition trials, the conditioned stimulus (i.e., activation of a sham electrode that can increase pain sensitivity, is paired to unconditioned high-pain stimuli (nocebo trials). During control trials of the acquisition phase, moderate-pain stimuli are paired to no sham electrode activation.
Behavioral: Extinction — During nocebo extinction, moderate pain stimulations are administered both after the administration of the conditioned stimulus (i.e., activation of the sham electrode) and the control stimulus (no activation of the sham electrode), in order to evoke nocebo responses to the sham hyperalgesic procedure.
Other: fMRI — In both arms of the study, BOLD response data will be collected with fMRI during the acquisition and extinction of nocebo effects on pain.
Drug: Placebo — Placebo control in oral form
  Arms: Baseline learning

SUMMARY:
Nocebo effects, negative responses to inert or active treatments which are putatively induced by negative outcome expectations, have been shown to play a significant role in pain perception. The underlying neurobiological mechanisms of these effects remain largely unexplored. The primary objective of this study is to test the role of N-methyl-D-aspartate (NMDA) receptor-dependent learning in an experimental model of conditioned nocebo effects on self-reported pain. Secondary objectives are to examine the role of the NMDA manipulation and related neural correlates during the acquisition and extinction of nocebo effects using statistical learning models. This study will utilize a placebo controlled, double-blind design with respect to the pharmacological administration of 80 mg D-Cycloserine (DCS), an NMDA agonist, or placebo. Validated conditioning and verbal suggestion (VS) paradigms will induce nocebo effects on pain in a random sample of 50 healthy adults. The primary endpoint of the study is the magnitude of the induced nocebo effect on pain measured as the difference between self-reported pain, between the first conditioned and control extinction trials. Secondary endpoints include the classification analysis of the Blood Oxygen Level Dependent (BOLD) responses of participants into pharmacological groups with multivariate pattern analysis. This study will be conducted at Leiden University and the Leiden University Medical Center (LUMC), The Netherlands.

DETAILED DESCRIPTION:
Main outcome variable:

- The magnitude of induced nocebo hyperalgesia is defined as the difference in pain ratings for the first nocebo trial compared to the first control trial of the extinction phase.

A significant difference here is assessed within the mixed model analysis of variance (ANOVA), comparing within-subjects differences for control and nocebo trials between DCS and placebo groups.

Time frame: On the day of the experimental session, during the extinction phase

Secondary outcome variables:

* The difference in BOLD response at a series of a priori ROIs between pharmacological groups during the acquisition of nocebo effects.
* The classification accuracy (into pharmacological groups), indicating that patterns of activation in the network of a priori ROIs form a model that can detect differences in neural activations during the acquisition of nocebo effects.
* The difference in BOLD response at a series of a priori ROIs between pharmacological groups during the extinction of nocebo effects.
* The classification accuracy (into pharmacological groups), indicating that patterns of activation in the network of a priori ROIs form a model that can detect differences in neural activations during the first trials of the extinction phase.
* The difference in BOLD response at a series of a priori ROIs between pain at baseline and nocebo-augmented pain.
* The classification accuracy, indicating that patterns of activation in the network of a priori ROIs form a model that can detect commonalities and differences in neural activations between the experience of pain at baseline and nocebo-augmented pain.
* The prediction accuracy, indicating that patterns of activation in the network of a priori ROIs form a model that can predict the magnitude of induced nocebo effects based on patterns of activations during the acquisition of nocebo effects.
* The moderation of the magnitude of induced nocebo effects in the first trials of the extinction phase by scores on the psychological questionnaires.

  0. Manipulation checks: Pain intensity responses during the acquisition phase To assess the effectiveness of the conditioning paradigm, pain ratings during acquisition will be analysed using a 2x1 mixed model ANOVA with group as a between-subjects factor (DCS, placebo), and pain intensity scores as a within-subjects, repeated measure with two levels (conditioned and unconditioned trials).

Effect of DCS on learning The Wechsler Memory Scale-Fourth Edition (WMS-IV) subtest Verbal Paired Associates will be used to assess whether DCS enhanced learning. A 2x1 mixed model ANOVA with group as the between-subjects factor and WMS-IV scores as the within-subjects repeated measure with two measurements, before administering DCS or placebo versus at two hours post-administration, before the beginning of the conditioning paradigm.

1. Primary hypothesis:

   The magnitude of the induced nocebo effect on pain is hypothesized to be larger in the DCS group relative to the placebo group. The magnitude of the nocebo effect is measured as the difference between self-reported pain on a Numeric Rating Scale (NRS) between the first conditioned and control extinction phase trials.
2. Secondary hypotheses:

   2.1. The magnitude of the conditioned nocebo effects still present after extinction is measured as the change from the average nocebo effect reported in the first trials of the extinction phase (after acquisition) and the average nocebo effect reported in last trials of the extinction phase (after extinction).

   2.2. DCS and placebo groups will be characterized by divergent neural activity across a set of a priori regions of interest (ROIs) during acquisition. ROI analysis of differences in BOLD responses will be performed on periaqueductal grey, (PAG), ventrolateral prefrontal cortex, (vlPFC), and dorsolateral prefrontal cortex (dlPFC), amygdala, anterior cingulate cortex (aCC), hippocampus, rostral ventromedial medulla (RVM), thalamus, insula.

   2.3 Multivariate pattern analysis (i.e., machine learning methods) will be used to investigate differences in BOLD responses during the acquisition of nocebo effects and thereby classify participants into pharmacological treatment groups (1) DCS, or 2) placebo) based on neural activity in the following ROIs: PAG, vlPFC, dlPFC, aCC, RVM, amygdala, thalamus, insula.

   2.4. DCS and placebo groups will be characterized by divergent BOLD responses across a set of a priori ROIs during extinction. ROI analysis for differences in BOLD responses between DCS and placebo groups will be performed on the following ROIs: PAG, vlPFC, dlPFC, aCC, RVM, amygdala, thalamus, insula.

   2.5 Multivariate pattern analysis will be used to investigate differences in BOLD responses during the extinction of nocebo effects and thereby classify participants into pharmacological treatment groups (1) DCS, or 2) placebo) based on neural activity in the following ROIs: PAG, vlPFC, dlPFC, aCC, RVM, amygdala, thalamus, insula.

   2.6. Pain and baseline, and nocebo augmented pain of a similar intensity will be characterized by divergent neural activations. Within the placebo group, ROI analysis for differences in BOLD responses between nocebo experiences and sensory experiences of pain based on BOLD responses in the following ROIs: PAG, vlPFC, dlPFC, aCC, RVM, amygdala, thalamus, insula.

   2.7. Pain and baseline, and nocebo augmented pain of a similar intensity will be characterized by divergent neural activations. Within the placebo group, multivariate pattern analysis will be used to investigate the differences in BOLD responses between nocebo experiences and sensory experiences of pain based on neural activity in the following ROIs: PAG, vlPFC, dlPFC, aCC, RVM, amygdala, thalamus, insula.

   . 2.8. Patterns of BOLD responses measured during the acquisition of nocebo effects in all pharmacological groups (1) DCS, or 2) placebo) at the previously listed ROIs, will predict the magnitude of nocebo effects on pain during extinction.
3. Questionnaires To assess the influence of psychological traits, questionnaires will also be included. These will include the Pain Catastrophizing Scale (PSC), Spielberger State Trait Anxiety Inventory (STAI), and the Body Vigilance Scale (BVS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 35 years
* Good understanding of the English language
* Normal or corrected to normal vision

Exclusion Criteria:

A potential participant who meets any of the following exclusion criteria will be excluded from participation in this study:

1. History of serious or chronic medical or psychiatric conditions (e.g., convulsions (epilepsy), cardiovascular problems, depression; careful and detailed screening will be carried out for both medical and psychiatric conditions)
2. History of chronic pain or itch conditions
3. Experiencing pain or itch of 1 or more on a 0-10 pain / itch NRS on the day of testing
4. Currently using antihistamines, analgesic medication, or itch-reducing medication (in the 24 hours prior to testing)
5. Use of psychotropic drugs (including recreational drugs such as cannabis and psychotropic prescription-medication; in the past month)
6. Currently being (or intending to become) pregnant, or currently breastfeeding, or planning to father a child in the next 3 months
7. Colour-blindness
8. Body Mass Index under 16 or over 30
9. Meeting any exclusion criteria in the fMRI examination questionnaire which would prohibit fMRI scanning.
10. Having too high of a threshold for pain (where high pain cannot be induced with temperatures lower than 49.5 °C).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants whose lived gender is male, will be included as male. Participants whose lived gender is female, will be included as female.
Enrollment: 53 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Magnitude of induced nocebo hyperalgesia | Through study completion, an average of 2 weeks
  is defined as the difference in pain numerical rating scale ratings (self-report, scale from 0 - no pain to 10 - worst pain imaginable) for the first nocebo trial compared to the first control trial of the extinction phase.
  A significant difference here is assessed within the mixed model ANOVA, comparing within-subjects differences for the control and nocebo trials between DCS and placebo groups

SECONDARY OUTCOMES:
The difference in blood-oxygen level dependent (BOLD) response at a series of a priori ROIs between pharmacological groups during the acquisition of nocebo effects. | Through study completion, an average of 2 weeks
  This will be measured via functional Magnetic Resonance Imaging assessing BOLD activations, for example hypo- and hyper- activation differences between the two pharmacological groups
The classification accuracy (into pharmacological groups), indicating that patterns of activation in the network of a priori ROIs form a model that can detect differences in neural activations during the acquisition of nocebo effects. | Through study completion, an average of 2 weeks
  This will be measured via functional Magnetic Resonance Imaging assessing BOLD activations, for example hypo and hyper activation differences between the two pharmacological groups
The difference in BOLD response at a series of a priori ROIs between pharmacological groups during the extinction of nocebo effects. | Through study completion, an average of 2 weeks
  This will be measured via functional Magnetic Resonance Imaging assessing BOLD activations, for example hypo and hyper activation differences between the two pharmacological groups
The classification accuracy (into pharmacological groups), indicating that patterns of BOLD activation in the network of a priori ROIs form a model that can detect differences in neural activations during the first trials of the extinction phase. | Through study completion, an average of 2 weeks
  This will be measured via functional Magnetic Resonance Imaging assessing BOLD activations, for example hypo and hyper activation differences between the two pharmacological groups
The difference in BOLD response at a series of a priori ROIs between pain at baseline and nocebo-augmented pain. | Through study completion, an average of 2 weeks
  This will be measured via functional Magnetic Resonance Imaging assessing BOLD activations, for example hypo and hyper activation differences between the two pharmacological groups
The classification accuracy, indicating that patterns of activation in the network of a priori ROIs form a model that can detect commonalities and differences in neural activations between the experience of pain at baseline and nocebo-augmented pain. | Through study completion, an average of 2 weeks
  This will be measured via functional Magnetic Resonance Imaging assessing BOLD activations, for example hypo and hyper activation differences between the two pharmacological groups
The prediction accuracy, indicating that patterns of activation in the network of a priori ROIs form a model that can predict the magnitude of induced nocebo effects based on patterns of activations during the acquisition of nocebo effects. | Through study completion, an average of 2 weeks
  This will be measured via functional Magnetic Resonance Imaging assessing BOLD activations, for example hypo and hyper activation differences between the two pharmacological groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrea WM Evers, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All data are collected pseudonymised thus no personal data are stored or shared. Consent forms are the only sources containing personal data and will not be shared, but are monitored by the department's Data Monitor.
  Supporting Information: Study Protocol; Statistical Analysis Plan (SAP); Analytic Code
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available immediately after publication of the study and will be retained for 15 years.
Access Criteria: Anonymized data can be shared with scientists in relevant fields for the purpose of future studies such as replication or meta-analysis (or with designated persons for monitoring purposes).